CLINICAL TRIAL: NCT02927925
Title: An Open Label, Phase 2 Study to Assess the Clinical Efficacy and Safety of Daratumumab in Patients With Relapsed or Refractory Natural Killer/T-Cell Lymphoma, Nasal Type
Brief Title: A Study to Assess the Clinical Efficacy and Safety of Daratumumab in Participants With Relapsed or Refractory Natural Killer/T-Cell Lymphoma (NKTCL), Nasal Type
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108237; 54767414NKT2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daratumumab (Experimental): Participants will receive daratumumab 16 milligram per kilogram (mg/kg) by intravenous (IV) infusion once weekly for 8 weeks, then every 2 weeks for 16 weeks, then every 4 weeks thereafter until study drug discontinuation due to progressive disease (PD), consent withdrawal or unacceptable toxicity.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Participants will receive daratumumab 16 mg/kg as intravenous infusion.

SUMMARY:
The purpose of this study is to assess the clinical efficacy and safety of daratumumab in relapsed or refractory natural killer/T-cell lymphomas (NKTCL).

ELIGIBILITY:
Inclusion Criteria:

* Documented as histologically confirmed extranodal natural killer/T-cell lymphomas (NK/T)-cell lymphoma, nasal type according to the World Health Organization (WHO) classification and the pathology report will be verified by the Sponsor
* Failed at least 1 line of chemotherapy and who, according to treating physician or investigator, is not candidate to receive other treatment modalities
* At least 1 measurable site of disease
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2 and life expectancy greater than or equal to (>=) 3 months

Exclusion Criteria:

* Received daratumumab or other antiCD38 therapies previously
* Previous allogenic stem cell transplant or autologous stem cell transplantation within 12 weeks before the first administration of the study drug
* Clinical symptoms of central nervous system involvement
* Known chronic obstructive pulmonary disease, known moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification
* Clinically significant cardiac disease, including:Myocardial infarction within 6 months before the first study agent administration, or unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association Class III-IV); Uncontrolled cardiac arrhythmia (Common Terminology Criteria for Adverse Events [CTCAE] [most recent version] Grade 3 or higher) or clinically significant ECG abnormalities; Screening 12-lead ECG showing a baseline QT interval as corrected QTc >470 msec
* Seropositive for human immunodeficiency virus
* Seropositive for hepatitis B or hepatitis C
* Abnormal laboratory values according to protocol defined parameters at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (17):
- China (5):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Beijing Cancer Hospital, Beijing
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - 1st Affiliated Hospital of Zhejiang University Medical College, Hangzhou
  - Ruijin Hospital, Shanghai Jiao Tong University, Shanghai
- Queen Mary Hospital, University of Hong Kong, Hong Kong, Hong Kong
- Singapore (2):
  - Singapore General Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (6):
  - National Cancer Center, Goyang-si
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Taiwan (3):
  - Changhua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Derived] Qing M, Zhou T, Perova T, Abraham Y, Sweeney C, Krevvata M, Zhang X, Qi M, Gao G, Kim TM, Yao M, Cho SG, Eom HS, Lim ST, Yeh SP, Kwong YL, Yoon DH, Kim JS, Kim WS, Zhou L, Attar R, Verona RI. Immune profiling of patients with extranodal natural killer/T cell lymphoma treated with daratumumab. Ann Hematol. 2024 Jun;103(6):1989-2001. doi: 10.1007/s00277-023-05603-w. Epub 2024 Jan 18. PMID 38233570
- [Derived] Huang H, Zhu J, Yao M, Kim TM, Yoon DH, Cho SG, Eom HS, Lim ST, Yeh SP, Song Y, Kwong YL, Kim JS, Jin J, Shi Y, Kim H, Qing M, Zhou T, Gao G, Dong Z, Qi M, Kim WS. Daratumumab monotherapy for patients with relapsed or refractory natural killer/T-cell lymphoma, nasal type: an open-label, single-arm, multicenter, phase 2 study. J Hematol Oncol. 2021 Feb 15;14(1):25. doi: 10.1186/s13045-020-01020-y. PMID 33588922

RESULTS

PARTICIPANT FLOW:
Groups:
- Daratumumab: Participants received daratumumab 16 milligrams per kilogram (mg/kg) as an intravenous (IV) infusion once weekly for 8 weeks, then every 2 weeks for 16 weeks, then every 4 weeks thereafter until study drug discontinuation due to progressive disease (PD), consent withdrawal or unacceptable toxicity (up to 392 Days).
Period: Overall Study
Arm/Group | Daratumumab
Started | 32
Completed | 0
Not Completed | 32
Not completed — Death | 16
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 11
Not completed — Other | 3
Not completed — Disease progression at clinical cutoff | 1

BASELINE CHARACTERISTICS:
Population: All treated analysis set included all the participants who have received at least one dose of study drug.
Arm/Group | Daratumumab
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 32
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  CHINA | 7
  HONG KONG | 1
  REPUBLIC OF KOREA | 17
  SINGAPORE | 2
  TAIWAN, PROVINCE OF CHINA | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response
Description: Overall response was defined as the percentage of participants who achieved complete response (CR) or partial response (PR) per Revised Criteria for Response Assessment of Hodgkin and non-Hodgkin lymphoma: LUGANO classification based on blinded independent central review (BICR). As per Revised Response Criteria for Malignant Lymphoma, Lymph node measurements were taken from Computed Tomography (CT), CT portion of the Positron Emission Tomography/Computed Tomography (PET/CT), where applicable. CR: complete disappearance of all evidence of disease; PR as a greater than (>) 50 percent (%) decrease in the sum of the products of the maximal perpendicular diameters of measured lesions (SPD) and no new sites.
Time Frame: Up to 2 years and 11 months
Population: All treated analysis set included all the participants who have received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 32
percentage of participants | 25.0 [11.5 to 43.4]

2. Secondary Outcome: Percentage of Participants With Complete Response (CR)
Description: CR was defined as the percentage of participants who achieved CR as per Revised Criteria for Response Assessment of Hodgkin and non-Hodgkin lymphoma: LUGANO classification based on BICR. CR was a complete disappearance of all evidence of disease.
Time Frame: Up to 2 years and 11 months
Population: All treated analysis set included all the participants who have received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 32
percentage of participants | 3.1 [0.08 to 16.22]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the duration from the date of the first daratumumab dose to the date of progression/relapse or death, whichever came first. Progressive disease (PD) was defined as any new lesion greater than (>) 1.5 centimeter (cm) in any axis or greater than or equal to (>=) 50 percent (%) increase in previously involved sites.
Time Frame: Up to 2 years and 11 months
Population: All treated analysis set included all the participants who have received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Daratumumab
Number analyzed (Participants) | 32
days | 53.0 [43.0 to 106.0]

4. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined as duration from the date of the initial documentation of a response to the date of first documented evidence of progressive disease (PD) (or relapse for participants who experienced CR). PD was defined as any new lesion >1.5 cm in any axis or >= 50% increase in previously involved sites.
Time Frame: Up to 2 years and 11 months
Population: All treated analysis set included all the participants who have received at least one dose of study drug and had CR or PR.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Daratumumab
Number analyzed (Participants) | 8
days | 55.0 [29.0 to 339.0]

5. Secondary Outcome: Time to Response
Description: Time to response was defined as the duration from the date of the first dose of daratumumab to the earliest date that a response (CR/PR based on BICR) is first documented. CR was defined as complete disappearance of all evidence of disease; PR as a greater than (>) 50 percent (%) decrease in the sum of the products of the maximal perpendicular diameters of measured lesions (SPD) and no new sites.
Time Frame: Up to 2 years and 11 months
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Daratumumab
Number analyzed (Participants) | 8
days | 52.0 [49 to 57]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from the date of the first daratumumab dose to the date of death.
Time Frame: Up to 2 years and 11 months
Population: All treated analysis set included all the participants who have received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Daratumumab
Number analyzed (Participants) | 32
days | 141.0 [94.0 to 235.0]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) as a Measure of Safety and Tolerability
Description: An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAE were defined as AEs with onset during the treatment period or that are a consequence of a pre-existing condition that has worsened since baseline.
Time Frame: Up to 2 years and 11 months
Population: All treated analysis set included all the participants who have received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 32
Participants | 26

8. Secondary Outcome: Number of Participants With Clinically Significant Change in Vital Signs
Description: Number of participants with clinically significant change in vital signs (blood pressure, temperature, pulse rate, and weight) was reported.
Time Frame: Up to 2 years and 11 months
Population: All treated analysis set included all the participants who have received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 32
Participants | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Number of participants with clinically significant ECG abnormalities were reported.
Time Frame: Up to 2 years and 11 months
Population: All treated analysis set included all the participants who have received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 32
Participants | 2

10. Secondary Outcome: Number of Participants With Clinically Significant Change in Physical Finding
Description: Number of participants with clinically significant change in physical finding was reported.
Time Frame: Up to 2 years and 11 months
Population: All treated analysis set included all the participants who have received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 32
Participants | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Change in Laboratory Parameters
Description: Number of participants with clinically significant change in hematology (WBC, hemoglobin, platelets, neutrophils, and lymphocytes) and biochemistry (alanine transaminase [ALT], aspartate transaminase [AST], sodium, potassium, bilirubin, alkaline phosphatase, calcium laboratory parameters were reported.
Time Frame: Up to 2 years and 11 months
Population: All treated analysis set included all the participants who have received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 32
Participants
  Hematology: WBC | 0
  Hematology: Hemoglobin | 0
  Hematology: Platelets | 0
  Hematology: Neutrophils | 0
  Hematology: Lymphocytes | 0
  Chemistry: ALT | 0
  Chemistry: AST | 0
  Chemistry: Sodium | 0
  Chemistry: Potassium | 0
  Chemistry: Bilirubin | 0
  Chemistry: Alkaline phosphatase | 0
  Chemistry: Calcium | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years and 11 months
Description: All treated analysis set included all the participants who have received at least one dose of study drug.
Arm/Group | Daratumumab
All-Cause Mortality (participants affected / at risk) | 21/32
Serious Adverse Events (participants affected / at risk) | 17/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daratumumab (N=32)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Periorbital Swelling (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Death (General disorders) | 1
Pyrexia (General disorders) | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 2
Epstein-Barr Virus Infection (Infections and infestations) | 1
Hepatitis Infectious Mononucleosis (Infections and infestations) | 1
Oral Candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Septic Shock (Infections and infestations) | 3
Skin Infection (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daratumumab (N=32)
Anaemia (Blood and lymphatic system disorders) | 9
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 7
Lymphopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Angina Pectoris (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Supraventricular Tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ear Discomfort (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Steroid Withdrawal Syndrome (Endocrine disorders) | 1
Cataract (Eye disorders) | 2
Diplopia (Eye disorders) | 1
Eye Swelling (Eye disorders) | 1
Periorbital Oedema (Eye disorders) | 1
Periorbital Swelling (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Vision Blurred (Eye disorders) | 3
Vitritis (Eye disorders) | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 4
Abdominal Pain (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 2
Anorectal Swelling (Gastrointestinal disorders) | 1
Aphthous Ulcer (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gingival Pain (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth Ulceration (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Proctalgia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 3
Chest Discomfort (General disorders) | 2
Chills (General disorders) | 8
Face Oedema (General disorders) | 2
Fatigue (General disorders) | 7
Generalised Oedema (General disorders) | 1
Influenza Like Illness (General disorders) | 2
Oedema (General disorders) | 1
Oedema Peripheral (General disorders) | 2
Pain (General disorders) | 4
Pyrexia (General disorders) | 20
Swelling Face (General disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Immunodeficiency (Immune system disorders) | 1
Eye Infection (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral Candidiasis (Infections and infestations) | 1
Oropharyngeal Candidiasis (Infections and infestations) | 1
Otitis Media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 3
Urinary Tract Infection (Infections and infestations) | 1
Limb Injury (Injury, poisoning and procedural complications) | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1
Alanine Aminotransferase Increased (Investigations) | 9
Aspartate Aminotransferase Increased (Investigations) | 8
Blood Alkaline Phosphatase Increased (Investigations) | 1
Blood Chloride Decreased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 2
Blood Lactate Dehydrogenase Increased (Investigations) | 1
C-Reactive Protein Increased (Investigations) | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1
Influenza B Virus Test Positive (Investigations) | 1
Interleukin Level Increased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 3
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck Pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraneoplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsions Local (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 8
Hypoaesthesia (Nervous system disorders) | 1
Limbic Encephalitis (Nervous system disorders) | 1
Lumbosacral Radiculopathy (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Haemoglobinuria (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 7
Skin Haemorrhage (Skin and subcutaneous tissue disorders) | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT02927925/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT02927925/SAP_001.pdf